CLINICAL TRIAL: NCT02658838
Title: The Application of Ticagrelor Combined With Low Molecular Weight Heparin During PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Zhao Jing Ye, Principal Investigator, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TLPCI
Record Dates: First submitted 2016-01-13; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-08

CONDITIONS: LOVASTATIN/TICAGRELOR [VA Drug Interaction]
MeSH Terms: interventions — Ticagrelor; Platelet Aggregation Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- full amount low molecular weight heparin (Experimental): Patients were treated with ticagrelor one year，After PCI， the patients are treated with full amount low molecular weight heparin until they leave hospital.
  Interventions: Drug: Ticagrelor; Drug: full amount low molecular weight heparin
- half amount low molecular weight heparin (Experimental): Patients were treated with ticagrelor one year，After PCI， the patients are treated with half amount low molecular weight heparin until they leave hospital.
  Interventions: Drug: Ticagrelor; Drug: half amount low molecular weight heparin
- No low molecular weight heparin (Experimental): Patients were treated with ticagrelor one year，After PCI， the patients are treated with no low molecular weight heparin.
  Interventions: Drug: Ticagrelor; Drug: No low molecular weight heparin

INTERVENTIONS:
Drug: Ticagrelor — Patients were treated with full amount low molecular weight heparin randomly after PCI,All patients are treated with ticagrelor one year.
  Other Names: Antiplatelet drugs
Drug: full amount low molecular weight heparin — Patients were treated with half amount low molecular weight heparin randomly after PCI,All patients are treated with ticagrelor one year.
  Other Names: Full amount enoxaparin
  Arms: full amount low molecular weight heparin
Drug: half amount low molecular weight heparin — Patients were treated with half amount low molecular weight heparin randomly after PCI,All patients are treated with ticagrelor one year.
  Other Names: Half amount enoxaparin
  Arms: half amount low molecular weight heparin
Drug: No low molecular weight heparin — Patients were treated with no low molecular weight heparin randomly after PCI,All patients are treated with ticagrelor one year.
  Other Names: No enoxaparin
  Arms: No low molecular weight heparin

SUMMARY:
The purpose of this study is to determine ticagrelor combining with low molecular weight heparin is effective and safe during PCI or not.

DETAILED DESCRIPTION:
Ticagrelor is a new drug compared with clopidogrel. It has a stronger antiplatelet capacity. After PCI，whether using low molecular weight heparin can make patients better prognosis or not, What's more，full amount or half amount low molecular weight heparin?, also investigators want to explore that whether it may lead to more bleeding events.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old and ≤75 years ;
2. unstable angina, non-ST segment elevation acute myocardial infarction, old myocardial infarction, or confirm the presence of myocardial ischemia;
3. voluntary participation in clinical trials, and informed consent;

Exclusion Criteria:

1. acute ST segment elevation myocardial infarction, stable angina pectoris;
2. aspirin allergy or resistance;
3. consolidated stroke, chronic obstructive pulmonary disease and other ticagrelor contraindications;
4. patients have coagulopathy;
5. can not be continued for one year with aspirin and treatment of dual antiplatelet ticagrelor;
6. can not complete revascularization;
7. NYHA ≥Ⅲ level or left ventricular ejection fraction <40%;
8. severe liver and kidney dysfunction (ALT and AST were more than three times the upper limit of normal, creatinine clearance less than 30ml / min-1.1.72m-2);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

SECONDARY OUTCOMES:
Nonfatal myocardial infarction | one year
  Patients occur acute myocardial infarction in a year，but it could not lead to die.
Non-fatal stroke | one year
  Patients occur stroke in a year，but it could not lead to die.
Revascularization again | one year
  Coronary arteries occur stenosis again in a year，the patients are treated with revascularization，including PCI and CABG.
Rehospitalization for ACS or heart failure | one year
  Patients are hospitalized again because of ACS or heart failure in a year.
Bleeding events | one year
  assessing the bleeding events according the TIMI grade.

CONTACTS AND LOCATIONS:
Overall Officials: jinghua Liu, Study Director — Beijing Anzhen hosipital
Locations (1):
- Beijing Anzhen Hosipital, Beijing, Beijing Municipality, China